CLINICAL TRIAL: NCT01226160
Title: Pilot Randomised Controlled Trial of Posturing Following Surgery for Full-thickness Macular Hole
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Moorfields Eye Hospital NHS Foundation Trust (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 06/Q0603/100/01
Record Dates: First submitted 2010-10-21; First posted 2010-10-22 (Estimated); Last update posted 2010-10-22 (Estimated); Status verified 2006-08

CONDITIONS: Full Thickness Macular Hole

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Face-down posturing group (Experimental): Postoperative face-down positioning for 10 days after surgery.
  Interventions: Procedure: Postoperative face-down posturing
- Non-posturing group (Active Comparator): avoid a face-up position for 10 days after surgery
  Interventions: Procedure: Postoperative non-posturing group

INTERVENTIONS:
Procedure: Postoperative face-down posturing — Postoperative face-down posturing for 10 days after surgery.
  Arms: Face-down posturing group
Procedure: Postoperative non-posturing group — avoid a face-up position only for 10 days after surgery
  Arms: Non-posturing group

SUMMARY:
This is a pilot randomised controlled trial (RCT) to investigate the effect of postoperative face-down positioning on the outcome of macular hole surgery.

ELIGIBILITY:
Inclusion Criteria:

* full thickness macular hole
* >16 years old

Exclusion Criteria:

* any history of previous intraocular surgery (including cataract surgery)
* history of ocular trauma
* history of visual loss greater than 1 year

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2005-01; Primary Completion 2010-02 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Anatomical closure of the macula hole assessed 6 weeks following surgery by ocular coherence tomography. | 6 weeks

SECONDARY OUTCOMES:
Visual acuity assessed 6 weeks following surgery by Snellen charts. | 6 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Moorfileld's Eye Hospital, London, London, United Kingdom